CLINICAL TRIAL: NCT06004258
Title: Effectiveness of the Painless Vaccination Protocol Versus Traditional Vaccination Methodology in Reducing Pain in Children Aged 2 Months to 14 Years. A Multicenter, Quasi-experimental (Non-randomized) Controlled Study
Brief Title: Reduction of Pain in Childhood Vaccination in the Primary Care Nurse Vaccination Consultation
Acronym: NoVacPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI_EFG_2022
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-06

CONDITIONS: Pain
Keywords: Vaccines; Pain Management; Primary Health Care; Infant; Child
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Quasi-experimental (non-randomized) controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental): Welcoming the child and his or her guardians Invite them to participate, explain the study, and collect informed consent Recording of vaccinations in the medical record Safety check-list and identification Structural and environmental adaptation of the office Decorated nursing uniforms Use of distracting and rewarding elements according to age Preparation of vaccines out of sight of children Apply antalgic measures according to age and preferences. If the skin is dirty, clean it with physiological saline solution. Administer vaccines from least painful to most painful Only cover the puncture site if there is bleeding. Give post-vaccination recommendations Measure pain before, during and after vaccination with validated scales according to age
  Interventions: Other: Painless Vaccination
- Control group (CG) (No Intervention): The "right 5+2" might be identified (patient, vaccine, interval, dose, route of administration, anatomical site, record) might be identified In infants, a non-pressing but secure breastfeeding position is recommended >3 years old: they sit on the tutor's lap, encouraging their collaboration to hold the child without compressing ensuring to avoid movements, and try to distract them 6-12 years old: they sit in the chair with the tutor sitting next to him/her and they are vaccinated asking for the child's collaboration. If necessary, they might be held to avoid movements Vaccines will be administered following The 2021 Vaccination Protocol Tutors will receive recommendations on adverse effects Queries might be solved The atmosphere of the immunization clinic is similar to the rest of the clinics in the health centre (white walls and no child decoration) The uniform used by the nurses is white and the vaccination techniques are the same as those previously used in these centres

INTERVENTIONS:
Other: Painless Vaccination — Structural adaptation of the vaccination areas and cozy decoration (colorful room, mobiles to hang on the ceiling) Nursing uniforms decorated with children's pictures Introduction of toys, stuffed animals, stamps and reward stickers, drawings and crayons, soothing music in the background
  Antalgic measures by age ranges:
  0-6M (FLACC scale) Breastfeed for two minutes if infant is breastfeeding Glucose 33% or 50% or if rotavirus vaccination, on mother's pacifier or gloved finger (non-nutritive sucking) Comfort between vaccinations 6-15M (FLACC scale) Position infant sitting on guardian's lap facing forward Distraction techniques: stuffed animals, toys, audiovisual devices 3-6Y (Wong-Baker scale) Involve child, explain Child sits on tutor's lap facing forward Distraction techniques: audiovisual devices, drawings 6-14Y (VAS scale)Always seated. Distraction method: audio-visual devices, breathing
  Arms: Intervention group (IG)

SUMMARY:
Non-randomized study with control group (CG) with the objective of analyzing the non-pharmacological analgesic efficacy of the "Painless Vaccine" protocol for the reduction of pain during vaccination in the population aged 2 months to 14 years participating in the experimental group (EG) versus traditional vaccination (CG).

DETAILED DESCRIPTION:
Administration of injectable vaccines is the most prevalent painful procedure in childhood-adolescence. Pain leads to decreased adherence to vaccination programs. There is scientific evidence on effective pharmacological and non-pharmacological interventions to reduce the pain associated with the act of vaccination. However, their application is scarce in our setting.

The aim of this study is to analyze the perception of pain during vaccination in the population aged 2 months to 14 years participating in the intervention group (IG) versus traditional vaccination (control group, CG).

Quasi-experimental study (non-randomized) with control group. The aforementioned population attending the primary care center for vaccination and whose guardian has given informed consent will be included. After training of the vaccination nurses of the GE and modifications of the environmental decoration, GE receives its vaccine in centers A and B; while in center C, the control group receives it in the traditional way.

The main outcome variables are: pain during and post-vaccination, and the independent variables: age of the child and guardian, sex, type of vaccine and antalgic measures, etc.

Descriptive, bivariate and logistic regression statistical analysis will be performed, following the application criteria of each test. IBM-SPSS-V26 software.

Approved by the Research Bioethics Committee. For the first time in our environment, an experimental study is developed in real practice on non-pharmacological analgesic measures in the process of infant vaccination. The reduction of pain perceived by the user will improve adherence to vaccination programs and other invasive techniques. The use of the "Painless Vaccination" protocol will favor the incorporation of evidence into clinical practice, as well as the adherence of professionals to low cost measures, for the humanization of child care. As a potential limitation, resistance to change by professionals is expected.

ELIGIBILITY:
Inclusion Criteria:

* Niñas/os de 2 meses a 14 años que acuden a las consultas del Programa de Vacunación infantil de Andalucía.
* Que al menos uno de sus padres/tutores haya firmado el consentimiento informado por representación del menor para participar en este estudio.
* Sin límite por población residencia.
* Que pertenezcan a las poblaciones de estudio (intervención y control).

Exclusion Criteria:

* No se han contemplado criterios de exclusión. Se tendrán en cuenta, si surgieran, casos especiales como: niños con TEA grado I-II-III (trastorno del espectro autista), niños con niveles de ansiedad muy altos condicionados por experiencias desagradables previas relacionadas con las agujas (hospitalizaciones, vías, …). Estos casos se serán valorados por el equipo coordinador

Ages: 2 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 495 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Pain immediately after injection | During the vaccination procedure
  It is expected to reduce by 20% the perception of pain during the vaccination act in the IG with respect to the CG. Defining the success of the interventions with an applicable Moderate-High pain measure from 0-3 (FLACCr Scale value 3-5 and 6), Wong-Baker Scale applicable from 3-7 years (Mild= 2; Moderate= 4-6) and Visual Analog Scale applicable from 6 years (Mild 0-2).
  We will proceed to distinguish the number of vaccines received by infants in the different visits/age group and the vaccines themselves, as some are more painful than others. The most painful vaccines: Triple Viral, Pneumococcal 13 and Human Papilloma Virus. The less painful vaccines: Hexavalent, Meningococcal C, and Tetravalent Meningococcal.
Pain before leaving the office | During the vaccination procedure
  It is expected to reduce by 20% the perception of pain during the vaccination act in the IG with respect to the CG. Defining the success of the interventions with an applicable Moderate-High pain measure from 0-3 (FLACCr Scale value 3-5 and 6), Wong-Baker Scale applicable from 3-7 years (Mild= 2; Moderate= 4-6) and Visual Analog Scale applicable from 6 years (Mild 0-2).
  We will proceed to distinguish the number of vaccines received by infants in the different visits/age group and the vaccines themselves, as some are more painful than others. The most painful vaccines: Triple Viral, Pneumococcal 13 and Human Papilloma Virus. The less painful vaccines: Hexavalent, Meningococcal C, and Tetravalent Meningococcal.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Franco García, BSN, Principal Investigator — Servicio Andaluz de Salud- Distrito Sanitario Aljarafe-Sevilla Norte
Locations (1):
- Distrito Sanitario Aljarafe-Sevilla Norte, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Centre for Disease Prevention and Control- Public Health Guidance. Revised 2016. Let´s talk about protection. Enchancing childhoot vaccination update.
- [Result] García Sánchez N, Merino Moína M, García Vera C, Lacarta García I, Carbonell Muñoz L, Pina Marqués B, et al. Alivio del dolor y el estrés al vacunar. Síntesis de la evidencia: recomendaciones del Comité Asesor de Vacunas de la AEP. Pediatría Atención Primaria. 2015;17(68):317-27.
- [Result] Birnie KA, Noel M, Chambers CT, Uman LS, Parker JA. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005179. doi: 10.1002/14651858.CD005179.pub4. PMID 30284240
- [Result] Taddio A, McMurtry CM, Shah V, Riddell RP, Chambers CT, Noel M, MacDonald NE, Rogers J, Bucci LM, Mousmanis P, Lang E, Halperin SA, Bowles S, Halpert C, Ipp M, Asmundson GJG, Rieder MJ, Robson K, Uleryk E, Antony MM, Dubey V, Hanrahan A, Lockett D, Scott J, Bleeker EV; HELPinKids&Adults. Reducing pain during vaccine injections: clinical practice guideline. CMAJ. 2015 Sep 22;187(13):975-982. doi: 10.1503/cmaj.150391. Epub 2015 Aug 24. No abstract available. PMID 26303247
- [Result] Centers for Diseases Control and Prevention. Epidemiology and Precention of Vaccine- Preventible Diseases.The Pink Book:Course text book- - 14.ª edición (2021) Epidemiología y Prevención de Enfermedades Prevenibles por Vacunación.
- [Result] Wallace AS, Mantel C, Mayers G, Mansoor O, Gindler JS, Hyde TB. Experiences with provider and parental attitudes and practices regarding the administration of multiple injections during infant vaccination visits: lessons for vaccine introduction. Vaccine. 2014 Sep 15;32(41):5301-10. doi: 10.1016/j.vaccine.2014.07.076. Epub 2014 Aug 1. PMID 25092632
- [Result] García Sánchez N, García SN, Hernández MA. Nuevos retos en vacunación. AEPap (ed.). Curso de Actualización Pediatría, 2017. Madrid: Lúa Ediciones 3.0; 2017. pp. 419-32
- [Result] Taddio A, Ilersich AF, Ilersich AN, Wells J. From the mouth of babes: Getting vaccinated doesn't have to hurt. Can J Infect Dis Med Microbiol. 2014 Jul;25(4):196-200. doi: 10.1155/2014/470261. PMID 25285123
- [Result] . Pardo Calderón HE, Yataco Chamorro RN. Efectividad de las técnicas no farmacológicas para el alivio del dolor postvacunal en los niños menores de 5 años [Internet]. Universidad Privada Norbert Wiener; 2018. Available from: http://repositorio.uwiener.edu.pe/bitstream/handle/123456789/2166/TITULO - Hilda Erika Pardo Calderón.pdf?sequence=1&isAllowed=y
- [Result] M. Ávila Carrasco a , L. Carbonell Muñoz a, A. Gómez Merino a, M. Méndez Perruca b, M.J. Rodríguez Besada b ¿Pueden los enfermeros de Atención Primaria contribuir en la disminución del dolor al vacunar? .Vacunas Volume 19, Issue 1, January-June 2018, Pages 8- 11
- [Result] Tomás Rojas J, Benítez Muñoz N, Menéndez Sotillos MI, Portellano Soriano MI, Caballero Aguilera F, Palomares Ojeda L. Vacunación en el Siglo XXI . Menos dolor , mejor ambiente , seguridad y confort. Garnata 91 [Internet]. 2020;22:1-7. Available from: http://www.ciberindex.com/index.php/g91/article/view/e202313/e202313
- [Result] Miranda C. Sanchez, et col. Tetanalgesia durante la vacunación de lactantes en atención primaria. Biblioteca Las Casa. http//www.index-f.com/lascasas/documentos/lc0874.php.2016.
- [Result] Harrison D, Reszel J, Bueno M, Sampson M, Shah VS, Taddio A, Larocque C, Turner L. Breastfeeding for procedural pain in infants beyond the neonatal period. Cochrane Database Syst Rev. 2016 Oct 28;10(10):CD011248. doi: 10.1002/14651858.CD011248.pub2. PMID 27792244
- [Result] Eden, L., et cols.. Minimizar el dolor durante las inyecciones de vacunación infantil: la mejora de la adherencia a los programas de vacunación. https://doi.org/10.2147/PHMT.S50510. 2014
- [Result] González-María E, Fuentelsaz-Gallego C, Moreno-Casbas T, Gil-Rubio P, Herreros-López P en nombre del grupo de trabajo de la G para el manejo del dolor en niños con cáncer. Guía de Práctica Clínica para el manejo del dolor en niños con cáncer [Internet]. 1a. Madrid, España: Investen; 2013. 142 p. Available from: http://www.criscancer.org
- [Result] Nieto Garcia A, Berbel Tornero O, Monleon Sancho J, Alberola-Rubio J, Lopez Rubio ME, Pico Sirvent L. [Evaluation of pain in children of 2, 4 and 6 months after the application of non-pharmacological analgesia methods during vaccination]. An Pediatr (Engl Ed). 2019 Aug;91(2):73-79. doi: 10.1016/j.anpedi.2018.10.002. Epub 2018 Nov 15. Spanish. PMID 30448108
- [Result] Kumar P, Sharma R, Rathour S, Karol S, Karol M. Effectiveness of various nonpharmacological analgesic methods in newborns. Clin Exp Pediatr. 2020 Jan;63(1):25-29. doi: 10.3345/kjp.2017.05841. Epub 2019 Aug 16. PMID 31431605
- [Result] Harrison D, Yamada J, Adams-Webber T, Ohlsson A, Beyene J, Stevens B. Sweet tasting solutions for reduction of needle-related procedural pain in children aged one to 16 years. Cochrane Database Syst Rev. 2015 May 5;2015(5):CD008408. doi: 10.1002/14651858.CD008408.pub3. PMID 25942496
- [Result] Bonnie Stevens1,2,3,4, Janet Yamada5, Arne Ohlsson6, Sarah Haliburton7, Allyson Shorkey7 Sacarosa para la analgesia de recién nacidos sometidos a procedimientos dolorosos Cochrane Database Syst Rev [Internet].2017 DOI: 10.1002/14651858.CD001069.pub5
- [Result] Taddio, A, Moshe, I. Vibhuti S. lIersich, L.Kikuta, Physical interventions and injection techniques to reduce pain by injection during routine immunizations in childhood.. 2016. https://www.ncbi.nlm.nih.gov/pubmed/19781436
- [Result] Psychological interventions with some evidence of benefit in children include: verbal distraction, video distraction, music distraction, and breathing with a toy.(1) Cochrane Data Base